CLINICAL TRIAL: NCT02691013
Title: The Impact of Ramelteon on Sleep and Delirium in Patients Who Undergo Pulmonary Thromboendarterectomy (PTE) Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Associate Professor, Pulmonary, Critical Care and Sleep Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 151294
Record Dates: First submitted 2015-12-28; First posted 2016-02-24 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Delirium; Sleep Deprivation
MeSH Terms: conditions — Delirium; Sleep Deprivation | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive a Placebo tablet every evening.
  Interventions: Drug: Placebo
- Ramelteon (Active Comparator): Patients will receive Ramelteon 8mg every evening.
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: Ramelteon
  Arms: Ramelteon
Drug: Placebo
  Arms: Placebo

SUMMARY:
Sleep deprivation is known to affect brain function but is often ignored in the sickest patients including those in the intensive care unit after major surgery. In these patients, the levels of melatonin can also be altered. Melatonin is a hormone secreted in the brain that maintains the body's sleep-wake, or circadian, cycle. The investigators want to test whether improving sleep quality affects the risk of developing confusion (delirium) in patients having clot removed from their lung (open heart surgery). In order to improve sleep quality, the investigators will conduct a study of Ramelteon, a medication that mimics the activity of melatonin and measure its effects on levels of melatonin and monitor sleep.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Thromboembolic Pulmonary Hypertension (CTEPH) who are admitted to UCSD for a planned PTE surgery.
* Age > 18 years

Exclusion Criteria:

* Pregnancy
* Cirrhosis of any etiology
* Current use of any atypical antipsychotic including Fluvoxamine (contra-indicated with Ramelteon)
* Any contraindication to EEG/Sleep recording
* Non-English speaking (who are unable to complete delirium questionnaires)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2022-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Owens, Principal Investigator — 8686577118

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Aama T, Brymer C, Gutmanis I, Woolmore-Goodwin SM, Esbaugh J, Dasgupta M. Melatonin decreases delirium in elderly patients: a randomized, placebo-controlled trial. Int J Geriatr Psychiatry. 2011 Jul;26(7):687-94. doi: 10.1002/gps.2582. Epub 2010 Sep 15. PMID 20845391
- [Background] Bellapart J, Boots R. Potential use of melatonin in sleep and delirium in the critically ill. Br J Anaesth. 2012 Apr;108(4):572-80. doi: 10.1093/bja/aes035. PMID 22419624
- [Background] Hatta K, Kishi Y, Wada K, Takeuchi T, Odawara T, Usui C, Nakamura H; DELIRIA-J Group. Preventive effects of ramelteon on delirium: a randomized placebo-controlled trial. JAMA Psychiatry. 2014 Apr;71(4):397-403. doi: 10.1001/jamapsychiatry.2013.3320. PMID 24554232
- [Derived] Jaiswal SJ, Bagsic SRS, Takata E, Kamdar BB, Ancoli-Israel S, Owens RL. Actigraphy-based sleep and activity measurements in intensive care unit patients randomized to ramelteon or placebo for delirium prevention. Sci Rep. 2023 Jan 26;13(1):1450. doi: 10.1038/s41598-023-28095-0. PMID 36702822
- [Derived] Jaiswal SJ, Vyas AD, Heisel AJ, Ackula H, Aggarwal A, Kim NH, Kerr KM, Madani M, Pretorius V, Auger WR, Fernandes TM, Malhotra A, Owens RL. Ramelteon for Prevention of Postoperative Delirium: A Randomized Controlled Trial in Patients Undergoing Elective Pulmonary Thromboendarterectomy. Crit Care Med. 2019 Dec;47(12):1751-1758. doi: 10.1097/CCM.0000000000004004. PMID 31567351

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients will receive a Placebo tablet every evening starting the night prior to the procedure for a maximum of 7 nights total.
  Placebo
- Ramelteon: Patients will receive Ramelteon 8mg every evening starting the night prior to the procedure for a maximum of 7 nights total.
  Ramelteon
Period: Overall Study
Arm/Group | Placebo | Ramelteon
Started | 61 | 59
Completed | 58 | 59
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: 120 enrolled. 3 participants withdrew prior to receiving any drug. Reporting the results of the 117 who were analyzed.
Groups:
- Placebo: Patients will receive a Placebo tablet every evening.
  Placebo
- Ramelteon: Patients will receive Ramelteon 8mg every evening.
  Ramelteon
- Total: Total of all reporting groups
Arm/Group | Placebo | Ramelteon | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 78
  >=65 years | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (15.8) | 58.1 (14.1) | 57.1 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 29 | 29 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 58 | 59 | 117

OUTCOME MEASURES:

1. Primary Outcome: Duration of Delirium
Description: Measured twice daily during the ICU stay using the Confusions Assessment Method instrument.
Time Frame: Twice daily for up to 10 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Placebo | Ramelteon
Number analyzed (Participants) | 58 | 59
hours | 16 [10 to 29] | 24 [14 to 37]

2. Primary Outcome: Total Duration of Sleep
Description: Participants wore an actigraphy device on their wrist for the duration of their ICU stay. This device continuously measures activity, and thus estimates sleep time.
Time Frame: Daily for up to 10 days
Population: Due to funding & logistical constraints, only a subset of subjects would've been able to do the electroencephalography (EEG) monitoring used for sleep assessment. Thus, Total Duration of Sleep was not measured and we focused on our a priori secondary outcome of incident delirium, a change made before the start of data collection or analysis.
Arm/Group | Placebo | Ramelteon
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Delirium
Description: Measured twice daily over the course of the ICU stay using the Confusion Assessment Method instrument
Time Frame: Twice daily for up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ramelteon
Number analyzed (Participants) | 58 | 59
Participants | 22 | 19

4. Secondary Outcome: Average Daily Critical Care Pain Observation Tool (CPOT)
Description: average daily pain level using the CPOT Participants can score from 0 to 6 on the CPOT scale, with 0 being no pain (calm, comfortable), and 6 representing significant pain/agitation.
Time Frame: 10 days
Reporting Status: Not Posted, anticipated posting 2021-12

5. Secondary Outcome: Length of Hospital Stay
Time Frame: Duration of hospital admission
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Ramelteon
Number analyzed (Participants) | 58 | 59
days | 12 [10 to 14] | 12 [10 to 16]

6. Secondary Outcome: Length of ICU Stay
Time Frame: Duration of hospital admission
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Ramelteon
Number analyzed (Participants) | 58 | 59
days | 4 [3 to 5] | 4 [3 to 6]

7. Secondary Outcome: Measures of Light Quality in the Patient's Room
Description: Light meter placed at bedside in patient room; this meter measured and recorded the light level in lux for ever minutes.
Time Frame: 3 days
Reporting Status: Not Posted, anticipated posting 2021-12

8. Secondary Outcome: Measures of the Sound Levels in the Patient's Room
Description: Sound meter was placed at bedside in each patient room. This meter measured and recorded the sound level in decibels every two seconds.
Time Frame: 3 days
Reporting Status: Not Posted, anticipated posting 2021-12

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Placebo | Ramelteon
All-Cause Mortality (participants affected / at risk) | 4/61 | 3/59
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/59
Other Adverse Events (participants affected / at risk) | 0/61 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT02691013/Prot_SAP_000.pdf